CLINICAL TRIAL: NCT04500002
Title: Adjuvant Isonicotinic Acid Hydrazide (INH) Pretreatment With Misoprostol for Induction of Abortion in First-trimester Missed Miscarriage: A Randomized Controlled Trial
Brief Title: Isonicotinic Acid Hydrazide (INH) Pretreatment With Misoprostol Versus Misoprostol Alone in Missed Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/354/3/19
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: IUCD Complication
MeSH Terms: interventions — Isoniazid; Misoprostol

STUDY DESIGN:
Intervention Model Description: double blind randomized parallel assign controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized parallel assign controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 tablets of isonicotinic acid hydrazide 300 mg will be given as single daily doses, 5 mg per day for two days at home and the third dose will be given on admission to hospital on day 3 and will be followed by vaginal misoprostol 800 mcg every three hours up to maximum three doses.
  Interventions: Drug: Isonicotinic Acid Hydrazide; Drug: Misoprostol
- Misoprostol (Active Comparator): Misoprostol Alone 800 mcg every three hours up to maximum three doses
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Isonicotinic Acid Hydrazide — total dose 900 mg per day for 3 days then Misoprosrol 800mcg will be given to all patients for induction of abortion
  Arms: INH
Drug: Misoprostol — Misoprosrol 800mcg will be given to all patients for induction of abortion

SUMMARY:
The primary endpoint was the success rate of adjuvant isonicotinic acid hydrazide (INH) and misoprostol versus misoprostol alone for medical termination of first-trimester pregnancy.

DETAILED DESCRIPTION:
According to the American college of obstetricians and gynecologists (2005), medical abortion is an acceptable alternative for surgical procedures in pregnant women with gestational age of less than 10 weeks based on the last menstrual period

Oral or vaginal misoprostol causes complete abortion in almost 85% of cases within seven days before the 12th week

Adjuvant isonicotinic acid hydrazide (INH) administration with misoprostol raises the rate of complete abortion

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 70 days gestation (<10 wks)
* Hemoglobin >10 g/dL.
* BMI between 18.5 kg/m2 and 30 kg/m2.
* Missed abortion

Exclusion Criteria:

* Molar pregnancy.
* Fibroid uterus.
* Uterine anomalies.
* Coagulopathy.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.
* Scared uterus (previous myomectomy, cesarean section, hysterectomy and ruptured uterus).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with gestational age of less than 10 week
Enrollment: 240 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
number of patients with complete abortion | 12 hours
  number of patients with complete abortion
time from induction to abortion | 12 hours
  time from induction to abortion

SECONDARY OUTCOMES:
number of the women will undergo dilatation and curettage after failed medical induction of abortion | 12 hours
  number of the women will undergo dilatation and curettage after failed medical induction of abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No